CLINICAL TRIAL: NCT07267195
Title: An In-Clinic Confinement Study to Assess Elements of Abuse Liability for Four Heated Tobacco Product (HTP) Consumables and Two HTP Devices
Brief Title: Abuse Liability for Four Heated Tobacco Product (HTP) Consumables and Two HTP Devices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD252501
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobacco (Experimental): Eligible participants will be randomized to one of 8 IP use sequences, such that one of the following IPs (A, B, C, D, E, F, G, N) will be used in each of the eight test sessions:
  Interventions: Other: Product A; Other: Product N; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G
- Menthol (Experimental): Eligible participants will be randomized to one of 8 IP use sequences, such that one of the following IPs (A, H, I, J, K, L, M, N) will be used in each of the eight test sessions:
  Interventions: Other: Product A; Other: Product N; Other: Product H; Other: Product I; Other: Product J; Other: Product K; Other: Product L; Other: Product M

INTERVENTIONS:
Other: Product A — Usual Brand filtered, non-menthol /menthol combustible cigarette
Other: Product N — Nicorette White Ice Mint 4 mg
Other: Product B — Signature Tobacco, Standard Mode, Device 1
  Arms: Tobacco
Other: Product C — Signature Tobacco, Boost Mode, Device 1
  Arms: Tobacco
Other: Product D — Roasted Tobacco, Standard Mode, Device 1
  Arms: Tobacco
Other: Product E — Signature Tobacco, Standard Mode, Device 2
  Arms: Tobacco
Other: Product F — Signature Tobacco, Boost Mode, Device 2
  Arms: Tobacco
Other: Product G — Roasted Tobacco, Standard Mode, Device 2
  Arms: Tobacco
Other: Product H — Fresh Menthol, Standard Mode, Device 1
  Arms: Menthol
Other: Product I — Fresh Menthol, Boost Mode, Device 1
  Arms: Menthol
Other: Product J — Menthol Capsule (Crushed), Standard Mode, Device 1
  Arms: Menthol
Other: Product K — Fresh Menthol, Standard Mode, Device 2
  Arms: Menthol
Other: Product L — Fresh Menthol, Boost Mode, Device 2
  Arms: Menthol
Other: Product M — Menthol Capsule (Crushed), Standard Mode, Device 2
  Arms: Menthol

SUMMARY:
This is a single-site, open-label, randomized, 8-way crossover study designed to evaluate elements of abuse liability (AL), including subjective effects and physiological measures (pharmacodynamics [PD]) and plasma nicotine uptake (pharmacokinetics [PK]), during and following ad libitum use of the study investigational products (IPs) by generally healthy adult smokers.

DETAILED DESCRIPTION:
Smokers who predominantly smoke non-menthol (Arm 1) and menthol (Arm 2) combustible cigarettes will be recruited into this AL study.

Potential participants will complete a pre-screening telephone interview. They will complete a Screening Visit to assess their eligibility within 45 days prior to check-in and enrollment.

Starting on Day -1, participants will check-in at the clinical site to complete procedures to re-confirm eligibility. Eligible participants will be enrolled and confined for 10 days. Participants will be randomized to one of 8 product use sequences using a Williams Design. Starting on Day 1, for each product use sequence, participants will evaluate one IP in each of eight separate daily test sessions, each following a 12-hour period of abstinence from all tobacco- and nicotine-containing products. At the end of all the test sessions each participant will have evaluated the six HTP IPs, including: three non-menthol IPs - arm 1; three menthol IPs - arm 2 using either a one-component (device 1) or two-component (device 2) HTP device. Participants will also evaluate both a high-AL comparator (participant's usual brand [UB] cigarette) and a low-AL comparator (a commercially available nicotine replacement therapy [NRT] gum [Nicorette® White Ice Mint, 4 mg nicotine; referred to hereafter as "NRT gum"]).

On Day 1 and continuing through Day 9, participants in both arms will participate in daily test sessions that will last for approximately 4 hours. Each test session will include collection of both PD (subjective and physiological) and PK measures, during and following IP use.

For both study arms, and approximately half a day prior to each respective Test Session, a Product Acclimation Period will allow participants ad libitum use of subsequent IP (~5 minutes for device1/device 2 IPs, ~30 minutes for NRT per use) at least twice as per randomized sequence for product familiarization prior to use in the next day's Test Session. Following each Product Acclimation Period, participants will have access to their UB cigarettes for ad libitum smoking until the 12-hour tobacco abstinence begins prior to each Test Session.

Safety will be monitored throughout the study by the Principal Investigator (PI) (or designee) by assessing adverse events (AEs), vital sign measurements, physical examinations (including an oral examination), and clinical laboratory tests.

The Medical Monitor will be available for consultation throughout the duration of the study and for any follow-ups after study discharge.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
* Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
* Smokes combustible, filtered, non-menthol (Arm 1 only) or menthol cigarettes (Arm 2 only), 83 mm to 100 mm in length as primary source of tobacco. Smokers who also use other tobacco products (e.g., ENDS, smokeless tobacco, HTPs) will not be excluded from study participation,
* Smokes an average of at least 10 cigarettes per day (CPD) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the PI.
* Agrees to smoke the same UB cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand and style currently smoked most frequently by the participant.
* Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening and at check-in (Day -1).
* Positive urine cotinine test (e.g., >200 ng/mL) via dipstick at Screening.
* Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes" (Heatherton et al., 1991).
* Willing to use the UB cigarette, Study IPs, and Nicorette® nicotine gum during the study period.
* Willing to abstain from tobacco and nicotine use for at least 12 hours prior to the start of each of four Test Sessions.
* Females must be willing to use a form of contraception acceptable to the PI from the time of signing the ICF until End-of-Study.
* Examples of acceptable means of birth control are, but not limited to:

  * Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral
  * oophorectomy, bilateral salpingectomy);
  * physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with
  * spermicide;
  * non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs
  * (e.g., Mirena or Kyleena);
  * vasectomized partner; or
  * post-menopausal and not on hormone replacement therapy
  * abstinence.
* Males must use an acceptable method of birth control from Day -1 "check-in" until the End-of-Study, unless they have had a vasectomy or are abstinent from heterosexual intercourse, or their female partner is not able to bear children.
* Agrees to an in-clinic confinement of 10 days (9 nights).
* BMI within 18.0 to 40.0 kg/m2, inclusive (minimum weight of at least 50.0 kg at Screening).

Exclusion Criteria:

* Individuals or their family members that have ongoing litigation with tobacco company(ies).
* Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
* History, presence of, or clinical laboratory test results indicating diabetes.
* Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion.
* History or presence of bleeding or clotting disorders.
* Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
* Systolic BP of > 160 mmHg or a diastolic BP of > 95 mmHg, measured after being seated for 5 minutes at Screening or at check-in Day -1.
* Weight of > 50.0 kg at Screening.
* Hemoglobin level is > 12.5 g/dL for females or > 13.0 g/dL for males at Screening.
* Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
* Has positive urine drug screen or alcohol test (urine or breath) at Screening or at Check-in to the Assessment Phase (Day -1), with the exception of positive results for tetrahydrocannabinol (THC). If positive for THC at check-in (Day -1), a cannabis intoxication evaluation will be performed, and inclusion will be at the discretion of the PI.
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
* Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), GLP-1 agonists (e.g., Mounjaro®, Ozempic®, Wegovy®), or lobelia extract within (≤) 30 days prior to signing the informed consent.
* Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous quit attempt within (≤) 30 days prior to signing the informed consent.
* Any use of daily aspirin (≥ 325 mg) or any use of other anticoagulants.
* Individuals ≥ 35 years of age currently using systemic, testosterone, estrogen-containing contraception or hormone replacement therapy.
* Whole blood donation or lost blood or blood products in excess of 500 mL within 8 weeks (≤ 56 days) prior to signing the informed consent and between Screening and check-in Day -1.
* Plasma donation within (≤) 7 days prior to signing the informed consent and between Screening and check-in Day -1.
* Employed by a tobacco or nicotine company, the study site, or handles raw, unpackaged tobacco- or nicotine-containing products as part of their job.
* Has used an investigational drug, device, biologic, or tobacco/nicotine product in a previous clinical study within 30 days or 5 times the half-life of the product (whichever is longer) prior to Screening.
* Drinks more than 21 servings of alcoholic beverages per week.
* Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AUECPL 3-240 | 3 minutes to 240 minutes
  area under the curve (AUEC) for PL (VAS score-versus-time) from 3 minutes to 240 minutes after the start of IP use
Emax PL | 240 minutes
  maximum effect (maximum PL VAS score after the start of IP use)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keyser, Study Director — Reynolds American

IPD SHARING:
Plan to Share IPD: No